CLINICAL TRIAL: NCT06648915
Title: Association of Lipoprotein(a) With Progression of Degenerative Aortic Valve Stenosis: Propensity-matched Study
Brief Title: Lipoprotein(a) and Progression of Aortic Stenosis
Status: Active, not recruiting | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Duk-Hyun Kang, Professor, Asan Medical Center
Other Study IDs: 2024-1209
Record Dates: First submitted 2024-10-15; First posted 2024-10-18 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Aortic Valve Stenosis; Lipoprotein(a)
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with mild to moderate AVS: Patients with measurements of Lp(a) and mild to moderate AVS
  Interventions: Diagnostic Test: Lipoprotein(a)

INTERVENTIONS:
Diagnostic Test: Lipoprotein(a) — Measurement of Lp(a) was performed at the time of entry to the registry. Lp(a) level was measured using immunenephelometric assay

SUMMARY:
This study is a prospective, observational, two arm parallel group, clinical study involving patients with measurements of Lp(a) and mild to moderate aortic stenosis. A total of 1381 patients underwent measurement of Lp(a) and had a diagnosis of mild to moderate, degenerative aortic stenosis between 2001 and 2020 in Asan Medical Center. Investigators selected a propensity-matched cohort of patients with Lp(a) >70 mg/dL and those with Lp(a) <30 mg/dL from the registry of patients with mild to moderate aortic stenosis to control risk factors for progression of aortic stenosis, and try to prospectively compare progression of aortic stenosis between the two groups (Lp(a) >70 mg/dL versus Lp(a) < 30 mg/dL). Investigators also evaluate interactions between Lp(a) groups and baseline clinical and echocardiographic variables for progression of aortic stenosis.

DETAILED DESCRIPTION:
Observational and genetic studies suggest that high levels of lipoprotein(a) (Lp[a]) increase the risk of calcific aortic valve stenosis (AVS). With the advancements of novel, specific therapies targeting Lp(a), there has been a growing need for clinical trials evaluating the effect of Lp(a) lowering in AVS. Requirement of longer follow-up time, selection of target populations and estimation of effect size are challenging issues for conducting clinical trials in AVS, and previous trials of statin therapy, which included patients with mild to moderate AVS, showed no significant effect of lowering LDL-cholesterol on the progression of AVS. Although post hoc analyses of previous statin trials showed that elevated levels of Lp(a) was associated with faster AVS progression, Lp(a) was associated with initiation but not with progression of AV calcification in a population-based study including 922 individuals. Because of a critical logistical challenge to randomized trials focusing the pre-calcific stages of AV disease, a clinical trial testing the progression of preexisting AVS is more feasible. The Lp(a)FRONTIERS CAVS trial (Assessing the Impact of Lipoprotein(a) Lowering with Pelacarsen (TQJ230) on the Progression of Calcific AVS; NCT05646381) will determine if pelacarsen can slow down the progression of AVS in patients with mild to moderate calcific AVS compared to placebo. To ensure adequate power to test the hypothesis of the ongoing Lp(a)FRONTIERS CAVS trial, it is important to estimate differences in progression of AS according to Lp(a) levels. However, such information is lacking and a well-designed prospective observational study is needed to directly compare progression of AS between the target population (patients with Lp(a) >70 mg/dL) of the Lp(a)FRONTIERS CAVS trial and control population (patients with mild to moderate AS and Lp(a) <30 mg/dL).

Investigators' prospective registry, started in 2001 at Asan Medical Center, has included all consecutive patients with measurements of Lp(a) and echocardiographic diagnosis of AVS. A total of 1381 patients underwent measurement of Lp(a) and had a diagnosis of mild to moderate, degenerative AVS between 2001 and 2020. Of the 1381 patients, 831 had Lp(a) level >70 mg/dL and 186 had Lp(a) level < 30 mg/dL. To reduce the effect of bias and potential confounding in this observational study, investigators performed rigorous adjustment for the differences in baseline characteristics using propensity-score matching. The propensity-score matched pairs were created by matching patients with Lp(a) >70 mg/dL and those with Lp(a) < 30 mg/dL in a 1:1 ratio. The primary cohort comprised 182 propensity-score matched pairs. The primary objective is to test the hypothesis that, compared with patients with Lp(a) < 30 mg/dL, those with Lp(a) >70 mg/dL have a faster progression of AVS in a propensity-matched cohort of patients with mild to moderate AVS. Investigators also try to evaluate interactions between Lp(a) groups and baseline clinical and echocardiographic variables for progression of AVS.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate degenerative AVS Aortic peak velocity greater than 2 m/s and smaller than 4 m/s
* LP(a) >70 mg/dL or <30 mg/dL
* Patients must provide written informed consent

Exclusion Criteria:

* Bicuspid AVS
* Rheumatic AVS
* Marked bradycardia, tachycardia or 2nd or 3rd degree AV block
* LV ejection fraction < 40%
* Hypertrophic or restrictive cardiomyopathy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent measurement of Lp(a) and had a diagnosis of mild to moderate, degenerative AVS between 2000 and 2020
Sampling Method: Non-Probability Sample
Enrollment: 364 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Annualized change in peak aortic jet velocity | From enrollment to the registry to performance of the last follow-up echocardiographic examination, assessed up to 36 months

SECONDARY OUTCOMES:
Annualized change in mean transvalvular gradient | From enrollment to the registry to performance of the last follow-up echocardiographic examination, assessed up to 36 months
Occurrence of the composite of cardiovascular events (progression to severe aortic stenosis, aortic valve replacement, or cardiovascular mortality) | From enrollment to the registry to performance of the last follow-up echocardiographic examination, assessed up to 36 months
Occurrence of all-cause mortality | From enrollment to the registry to performance of the last follow-up echocardiographic examination, assessed up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Duk-Hyun Kang, MD. PhD., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No